CLINICAL TRIAL: NCT05847608
Title: Concussion and Omega-3s - New Consideration for the Therapeutic Use of Nutritional Supplements in Adolescents
Brief Title: Omega-3 Treatment for Concussion in Adolescents
Acronym: CONCUSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2023:018
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-04

CONDITIONS: Concussion, Mild
Keywords: Omega-3
MeSH Terms: conditions — Brain Concussion | interventions — Docosahexaenoic Acids; Eicosapentaenoic Acid; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 Supplementation (Experimental): This groups will supplement their regular diet with 1 tsp of fish oil containing 1.5 grams combined omega-3 fatty acid (EPA/DHA) supplement in liquid form on a daily basis until they are recovered or have been enrolled for 6 weeks.
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): This group will supplement their regular diet with 1 tsp olive oil in liquid form on a daily basis until they are recovered or have been enrolled for 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — Daily consumption of 500 mg DHA and 750 mg EPA in liquid form
  Other Names: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)
  Arms: Omega-3 Supplementation
Dietary Supplement: Placebo — Oleic Acid, Linoleic Acid
  Other Names: Olive Oil
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test omega-3 fatty acid supplementation as a treatment in adolescents with a concussion. The main questions it aims to answer are:

* Does supplementing with omega-3 fatty acids improve time to recovery following sport related concussion.
* Does supplementing with omega-3 fatty acids improve health related quality of life following concussion.
* Does supplementing with omega-3 fatty acids change post-concussion symptoms following concussion.
* Does supplementing with omega-3 fatty acids change saliva concentrations of interleukin-6 following concussion.
* Does supplementing with omega-3 fatty acids change saliva concentrations of cortisol following concussion.

Participants will be randomized to receive either an omega-3 supplement or placebo after they have been diagnosed with a concussion. Researchers will compare the omega-3 supplement group and placebo group to see if omega-3 fatty acids, consumed as a treatment, can improve time to recovery, health related quality of life and symptom burden, and whether omega-3 fatty acids alter interleukin-6 and cortisol concentrations in saliva following a concussion.

DETAILED DESCRIPTION:
Following mild traumatic brain injury, a neurometabolic cascade occurs with concurrent neuronal disruptions, metabolic changes, excitotoxicity, and changes in cerebral blood flow. Omega-3 fatty acids have been postulated as a possible nutritional supplement which could aid in recovery following a concussion. The omega-3 fatty acids docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) are derived from alpha-linolenic acid (ALA) which is an essential fatty acid. DHA is present at high concentrations in neuronal cells and contributes to the regulation of cell membranes, neurotransmitter release, neurogenesis, and neuroinflammation. EPA is converted to E-series resolvins which act in an anti-inflammatory manner.

Pre-clinical research supports the potential benefits of omega-3 fatty acids following a TBI. There has recently been one pilot study in human adolescents which also supports the need for large randomized controlled trials to fully understand the impact omega-3 fatty acids may have on recovery following concussion. The current evidence suggests that omega-3 supplementation may ameliorate neuroinflammation and neuronal apoptosis, and decrease reactive oxygen species associated with TBI. It has been suggested that following TBI, omega-3 supplementation may improve neural plasticity and signaling related molecules which can improve cognitive function following TBI.

Based on these previous mentioned studies it appears that omega-3 fatty acids could potentially benefit those recovering from a concussion. However, to date there have not been any appropriately powered randomized controlled trials evaluating the efficacy of omega-3 supplementation following sport related concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form;
2. State their willingness to comply with all study procedures and availability for the duration of the study;
3. Be between 14 and 17 years of age or older;
4. Meet the diagnostic criteria of a concussion set forth by the Consensus Statement on Concussion in Sport 5th Annual Conference of Concussion in Sport, 2017 as determined by the treating physician;
5. Present with a sport related concussion within 7 days from injury; and
6. Assigned a Glasgow coma scale (GCS) score = 15.

Exclusion Criteria:

1. Patients with a history of moderate or severe traumatic brain injury, epilepsy, or stroke;
2. Patients who have been diagnosed with a skull fracture, traumatic subarachnoid hemorrhage, subdural hematoma, epidural hematoma, intraparenchymal hemorrhage or cerebral contusion on previous neuro-imaging studies;
3. Pregnant patients;
4. Patients with a GCS score less than or equal to 14;
5. Patients for whom parental/guardian consent cannot be obtained;
6. Patients who have consumed an omega-3 fatty acid containing supplement within the past month;
7. Patients with a fish or shell fish allergy.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery | Maximum of 6 weeks
  Time to clinical recovery will be determined by the patients treating physician. This will be defined as: 1) symptoms have returned to baseline or resolved, 2) normal medical examination, 3) tolerating school full-time without symptoms, and 4) tolerating appropriate return to play steps and are cleared to participate in full sport activities.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (Version 4.0) Teen Report | Maximum of 6 weeks
  Participants will complete the paediatric quality of life inventory (https://www.pedsql.org/index.html) each week until the participant is determined to be clinically recovered or have not recovered by 6 weeks. Scale minimum score is 0 and maximum is 52. Higher scores mean worse outcome.
Pediatric Quality of Life Inventory (Version 4.0) Parents Report | Maximum of 6 weeks
  Parent/guardian will complete the paediatric quality of life inventory (https://www.pedsql.org/index.html) each week until the participant is determined to be clinically recovered or have not recovered by 6 weeks. Scale minimum score is 0 and maximum is 52. Higher scores mean worse outcome.
Sport Concussion Assessment Tool - 5 Symptom Evaluation | Maximum of 6 weeks
  Participants will report their symptoms using the post-concussion symptom scale ((PCSS; version from the Sport Concussion Assessment Tool-5) each week until they are determined to be clinically recovered or have not recovered by 6 weeks. Scale minimum score is 0 and maximum is 132. Higher scores mean worse outcome.
Interleukin-6 | Maximum of 6 weeks
  Interleukin-6 will be analyzed via enzyme-linked immunosorbent assay (ELISA) to determine changes in inflammatory status.
Cortisol | Maximum of 6 weeks
  Cortisol will be analyzed via enzyme-linked immunosorbent assay (ELISA) to determine changes in stress status.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cornish, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Applied Research Centre, Faculty of Kinesiology, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No